CLINICAL TRIAL: NCT03213782
Title: Effect of Nature Based Sounds' Intervention on Agitation and Anxiety of Patients Admitted in Intensive Care Units of MMIMS&R Hospital, Mullana, Ambala
Brief Title: Effect of Nature Based Sounds' Intervention on Agitation and Anxiety of Patients Admitted in Intensive Care Units.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Amandeep kaur, Principal Investigator, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200014
Record Dates: First submitted 2017-06-27; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Agitated; State, Acute Reaction to Stress; Anxiety
Keywords: Nature Based Sounds; Agitation; Anxiety; Patients; Intensive Care Units
MeSH Terms: conditions — Psychomotor Agitation; Stress Disorders, Traumatic, Acute; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Nature based sounds are administered via head phones continuously for 20 minutes.
  Interventions: Other: Nature based sounds
- Control group (No Intervention): Usual routine care was continued

INTERVENTIONS:
Other: Nature based sounds — Nature based sound was administered to the experimental group with head phones for continuously 20minutes. Posttest was done by continuously 30 minute observation after administration of nature based sound with the same tools.
  Arms: Experimental group

SUMMARY:
Effect of nature based sounds' intervention on Agitation and Anxiety of patients admitted in Intensive Care Units of MMIMS&R Hospital, Mullana, Ambala

DETAILED DESCRIPTION:
INTRODUCTION: Continue stay in ICU can lead to sleep disturbances and poor stress management that may result in client's inability to adjust with the situations and use of medical support. This experience may lead to increase agitation, anxiety as well as physiological stress of client, decrease comfort level and increase recovery time as well as hospital stay. There has been great emphasis on non-pharmacological methods that decrease anxiety and stress since they are very appropriate and affordable.

OBJECTIVES: The objective of the study was to assess the effect of Nature Based Sounds on Agitation and Anxiety of patients admitted in Intensive Care Units.

METHODOLOGY: A Randomized Controlled Trial with pretest posttest control group design was used. Sixty patients from Surgical Intensive care unit and were selected conveniently and randomly assigned into experimental and control group using lottery method. Data was collected by Agitation Behavior Assessment Scale and Beck Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study.
2. In age group of 18 -75 years.

Exclusion Criteria:

1. Patients who were not having agitated behavior, normal anxiety and normal physiologic stress scores.
2. Patients who were taking anti-hypertensive drugs, anti-depressants drugs and sedatives.
3. Who could not response verbally or non-verbally in response to Sample Characteristics Performa and Beck Anxiety Inventory.
4. Patients who were having psychiatric or neurological illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-01-07 (Actual); Study Completion 2017-01-07 (Actual)

PRIMARY OUTCOMES:
Agitation assessed with the Agitation Behavior Assessment Scale | 8-10 minutes
  Agitation Behavior Assessment Scale
  A Score of 14 = absent: the behavior is not present.
  15-28= low degree.
  29-42= Moderate degree.
  43-56= Extreme degree.

CONTACTS AND LOCATIONS:
Overall Officials: Mrs. Vinay Kumari, Msc. Nursing, Study Director — MM University, Mullana, Ambala, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woods JC, Mion LC, Connor JT, Viray F, Jahan L, Huber C, McHugh R, Gonzales JP, Stoller JK, Arroliga AC. Severe agitation among ventilated medical intensive care unit patients: frequency, characteristics and outcomes. Intensive Care Med. 2004 Jun;30(6):1066-72. doi: 10.1007/s00134-004-2193-9. Epub 2004 Feb 14. PMID 14966671
- [Background] Jaber S, Chanques G, Altairac C, Sebbane M, Vergne C, Perrigault PF, Eledjam JJ. A prospective study of agitation in a medical-surgical ICU: incidence, risk factors, and outcomes. Chest. 2005 Oct;128(4):2749-57. doi: 10.1378/chest.128.4.2749. PMID 16236951
- [Background] Gullich I, Ramos AB, Zan TR, Scherer C, Mendoza-Sassi RA. Prevalence of anxiety in patients admitted to a university hospital in southern Brazil and associated factors. Rev Bras Epidemiol. 2013 Sep;16(3):644-57. doi: 10.1590/s1415-790x2013000300009. English, Portuguese. PMID 24896278
- [Result] Saadatmand V, Rejeh N, Heravi-Karimooi M, Tadrisi SD, Zayeri F, Vaismoradi M, Jasper M. Effect of nature-based sounds' intervention on agitation, anxiety, and stress in patients under mechanical ventilator support: a randomised controlled trial. Int J Nurs Stud. 2013 Jul;50(7):895-904. doi: 10.1016/j.ijnurstu.2012.11.018. Epub 2012 Dec 14. PMID 23245705
- [Result] Aghaie B, Rejeh N, Heravi-Karimooi M, Ebadi A, Moradian ST, Vaismoradi M, Jasper M. Effect of nature-based sound therapy on agitation and anxiety in coronary artery bypass graft patients during the weaning of mechanical ventilation: A randomised clinical trial. Int J Nurs Stud. 2014 Apr;51(4):526-38. doi: 10.1016/j.ijnurstu.2013.08.003. Epub 2013 Aug 29. PMID 24035670
- [Result] Garland A, Olafson K, Ramsey CD, Yogendran M, Fransoo R. Epidemiology of critically ill patients in intensive care units: a population-based observational study. Crit Care. 2013 Sep 30;17(5):R212. doi: 10.1186/cc13026. PMID 24079640